CLINICAL TRIAL: NCT06354465
Title: Injectable Extended-Release Buprenorphine (XR-B) in a Correctional Setting: Qualitative Interviews
Status: Recruiting | Type: Observational
Sponsor: Lifespan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Justin Berk, Assistant Professor, Lifespan
Other Study IDs: IRB1967355; K23DA055695 (NIH)
Record Dates: First submitted 2024-03-31; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Opioid Use Disorder; Criminal Justice; Treatment Adherence and Compliance
Keywords: addiction; criminal justice; Medications for opioid use disorder
MeSH Terms: conditions — Opioid-Related Disorders; Treatment Adherence and Compliance; Behavior, Addictive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Incarcerated Individuals: Incarcerated individuals will be recruited across the Rhode Island Department of Corrections (RIDOC)facility during the required group sessions for treatment; this is consistent with previous NIH-funded studies at RIDOC. The interviews will be described and participants will be able to sign up confidentially. Participants who are eligible for Medications for Opioid Use Disorder (MOUD) but decide not to pursue treatment will still be interviewed to provide better understanding of the key factors that drive program participation. These individuals can be recruited through routine clinical care by addiction medicine providers. Every precaution will be taken to ensure confidentiality and protection of all participants.
- Stakeholders: Organizational stakeholders (clinicians, Wardens, leadership and/or other staff) will be recruited through snowball sampling. I will individually approach leaders of each facility to recruit correctional individuals interested in participating and will also allow participants to confidentially sign up at administrative meetings related to Medication for Addiction Treatment (MAT).

SUMMARY:
This qualitative study investigates the potential benefits and challenges of using a once-a-month injectable medication, known as extended-release buprenorphine (XR-B), to treat individuals with opioid use disorder (OUD) within a correctional setting. The research aims to understand if XR-B can be a feasible and effective alternative to the standard daily treatment and to identify which groups within the prison population may benefit the most from this treatment. In-depth interviews are conducted with incarcerated individuals and relevant stakeholders.

ELIGIBILITY:
Incarcerated individuals, inclusion criteria:

* English speaking
* Over the age of 18
* Diagnosed with opioid use disorder

Incarcerated individuals, Exclusion Criteria:

- Diagnosed with "Severe, Persistent, Mental Illness (SPMI)" Rationale for Exclusion: These individuals suffer from severe mental health disease and therefore warrant greater protection, have greater risk for coercion, and offer insights to severe co-diagnosis treatment that, while important, remain outside the scope of general MAT implementation.

Organizational Stakeholders, Inclusion Criteria:

- Employed or contracted by Rhode Island Department of Corrections (for organizational staff interviews) and involved with the Medication for Addiction Treatment (MAT) program

Organizational Stakeholders, Exclusion Criteria:

- If not permitted by their organizational union to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Incarcerated individuals include participants in the RIDOC MOUD program.
  Organizational stakeholders inlcude clinicians, Wardens, leadership and/or other staff involved in the MOUD program.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative Transcripts | 1 year
  A directed content analysis will identify key themes in structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Justin Berk, MD, Principal Investigator — Lifespan
Locations (1):
- Rhode Island Department of Corrections, Cranston, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided
Given the sensitivity of data, some individual data may be censored but will be available to other researchers in aggregate.

DOCUMENTS (2):
  • Study Protocol (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT06354465/Prot_000.pdf
  • Informed Consent Form (2023-01-07): https://cdn.clinicaltrials.gov/large-docs/65/NCT06354465/ICF_001.pdf